CLINICAL TRIAL: NCT05251792
Title: Study on the Relationship Between Macular Pigment Optical Density and Primary Angle-closure Disease
Brief Title: Macular Pigment Optical Density in Primary Angle-closure Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020KYPJ82
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-02

CONDITIONS: Glaucoma; Glaucoma, Angle-Closure; Macular Pigment Optical Density
Keywords: Glaucoma, Angle-Closure; PACD-Primary Angle Closure Disease; Macular Pigment Optical Density
MeSH Terms: conditions — Glaucoma; Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Angle Clousure Diseases Eyes: Over 40 years old, regardless of gender. Patients diagnosed with PACD (PACG or PAC or PACS) with phakic eyes. Peripheral iridectomy or trabeculectomy, more than 3 months after operation.
  Interventions: Other: Ocular examination
- Matched Eyes: Healthy population matched by sex and age.
  Interventions: Other: Ocular examination

INTERVENTIONS:
Other: Ocular examination — All participants underwent a detailed examination, including visual acuity, slit lamp biomicroscopy, direct ophthalmoscopy, optometry noncontact tonometry,MPOD measurement and optical coherence tomography (OCT) measurement

SUMMARY:
Glaucoma is the leading cause of irreversible blindness in the world, and primary angle-closure glaucoma (PACG) is the most important type of glaucoma in Asia. Primary angle closure disease (PACD) is a group of diseases related to PACG, and the pathogenesis is still unclear. Macular pigment has the functions of filtering short-wavelength waves and anti-oxidation, which are related to visual function. Previous studies have found that the macular pigment density (MPOD) is significantly reduced in primary open-angle glaucoma. This project uses the single-wavelength reflection method to measure MPOD, observes the characteristics of PACD and the normal control group's changes in retinal MPOD, and explains the relationship between PACD's MPOD changes and angle-closure glaucoma optic nerve damage

DETAILED DESCRIPTION:
Observation index： Visual acuity，Intraocular pressure，Ophthalmoscope，MPOD，Visual field and OCT.

Inspection parameters of OCT：

1. Retinal nerve fiber layer thickness
2. Ganglion cell complex thickness
3. Mean thickness of the central retina
4. Mean defect

ELIGIBILITY:
Inclusion Criteria:

* Experimental group：
* (1) According to the diagnostic criteria of PACD
* (2)History of peripheral iridectomy or trabeculectomy
* (3)Over 40
* (4)Phakic eyes
* (5)Intraocular pressure is less than 21mmhg, more than one week
* (6)Eyes with clear optical media.
* Control group：
* (1)No history of glaucoma and other eye diseases
* (2)Phakic eyes
* (3)Over 40
* (4)Intraocular pressure10~21mmHg

Exclusion Criteria:

* (1)History of corneal diseases
* (2)History of eye tumor or other ophthalmic surgery
* (3)Cataract
* (4)Taking supplements containing lutein within 6 months
* (5)Snellen's visual acuity was less than 6 / 20，the diopter is beyond ± 6 degrees

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients >=40 years old PACD
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Macular Pigment Optical Density（MPOD）Measurement | 3 months after surgery
  A one-wavelength fundus reflectance method (Visucam 200; Carl Zeiss Meditec) was used for the detection of MPOD as previously described. The right or left eye was randomly selected for measurement. The parameters and profiles of MPOD in a 7-degree eccentricity that corresponded to a 4 mm diameter were evaluated and output. Parameters included max and mean optical density (OD), volume, and area. MaxOD and MeanOD with units "d.u." (initial of density units) were used for the analyses.
Retinal nerve fiber layer thickness | 3 months after surgery
  Detection by optical coherence tomography (OCT). Circumpapillary RNFL scans were obtained using the standard 3.4 mm 12-degree circumpapillary nerve fiber layer scan protocol.We recorded superior, inferior, nasal, temporal, and total RNFL thickness.
Ganglion cell complex (GCC)thickness | 3 months after surgery
  Detection by optical coherence tomography (OCT). The distance from the internal limiting membrane and outer edge of the outer plexiform layer was defined as GCC thickness.
Mean central retina thickness | 3 months after surgery
  Detection by optical coherence tomography (OCT). CRT thickness was defined as distance between the internal limiting membrane and the inner edge of the retinal pigment epithelium.
Mean outer retinal thickness | 3 months after surgery
  Outer retinal (OR) thickness was calculated by subtracting GCC thickness from CRT.
Visual Field Test | 3 months after surgery
  The visual field test uses the 30-2 Threshold Test on the Humphrey Visual Field Analyzer.According to the mean deviation (MD) values generated by the software, three groups of disease severity were classified: the mild group with MD > -6 dB, the moderate group with MD between -6 and -12 dB, and the severe group with MD < -12 dB

SECONDARY OUTCOMES:
Visual acuity | 3 months after surgery
  Use Snellen visual acuity chart to measure naked eye vision and best corrected vision
Intraocular pressure | 3 months after surgery
  Using non-contact tonometer (NCT) measuring intraocular pressure
Cup/ Disk ( C/ D） | 3 months after surgery
  determine the cup to disc ratio by ophthalmoscope

CONTACTS AND LOCATIONS:
Overall Officials: Chengguo Zuo, Study Director — Zhognshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) needed to be keep security.